CLINICAL TRIAL: NCT04944680
Title: Effects of Transcranial Direct Current Stimulation and Motor Imagery for the Recovery of Upper Limb Function of Stroke Patients
Brief Title: Dual Channel Rehabilitation Technology Promotes Rapid Recovery of Upper Limbs After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Xing Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Ran Li, Doctor Li, Fu Xing Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021FXHEC-KSKY002
Record Dates: First submitted 2021-06-12; First posted 2021-06-29 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Stroke; Upper Extremity Dysfunction; Transcranial Direct Current Stimulation; Image, Body
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The four parallel groups are as follows: control group, Transcranial Direct Current Stimulation group, motor imagery group, Transcranial Direct Current Stimulation and motor imagery group. Patients are randomly assigned to each group with block randomization.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Because of the different therapies, it is not possible to mask the participant. It was possible to mask the group allocation for routine rehabilitation therapist. However, the difference is obvious between Transcranial Direct Current Stimulation and motor imagery. Outcome measure is conducted by a physician who is blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): Stroke patients accept the traditional rehabilitation alone.
- Transcranial Direct Current Stimulation group (Active Comparator): Stroke patients accept the Transcranial Direct Current Stimulation alone.
  Interventions: Behavioral: Transcranial Direct Current Stimulation therapy
- Motor imagery group (Active Comparator): Stroke patients do the motor imagery alone.
  Interventions: Behavioral: Motor imagery therapy
- Transcranial Direct Current Stimulation and motor imagery group (Experimental): Stroke patients accept the Transcranial Direct Current Stimulation and do the motor imagery at the same time.
  Interventions: Behavioral: Transcranial Direct Current Stimulation and motor imagery therapy

INTERVENTIONS:
Behavioral: Transcranial Direct Current Stimulation therapy — Transcranial Direct Current Stimulation with two saline-soaked electrodes (5cm x 7cm) is applied by our occupational therapist. The anode is placed on the ipsilesional primary motor cortex (C3/C4). The cathode is placed on the contralesional shoulder. The current is 1.5 milliampere and lasts 20 minutes.
  Arms: Transcranial Direct Current Stimulation group
Behavioral: Motor imagery therapy — Stroke patients are asked to watch a video about the upper extremity movement. The video lasts 20 minutes. The contents are as follows: the patients are asked to relax the muscles for the first 2 minutes; the action refers to shoulder flexion and extension, elbow flexion and extension, forearm pronation and supination, wrist flexion and extension, finger flexion and extension, and corresponding daily functional activities for 16min; the patients are asked to relax their mind and body for the last 2 minutes.
  Arms: Motor imagery group
Behavioral: Transcranial Direct Current Stimulation and motor imagery therapy — The treatment parameters are the same as the above. It should be emphasized that the participants sit and perform the motor imagery task while receiving Transcranial Direct Current Stimulation.
  Arms: Transcranial Direct Current Stimulation and motor imagery group

SUMMARY:
The injury and remodeling mechanism about upper extremity motor network after stroke is not clear. There are few studies on the motor network covering cortex, white matter and blood perfusion at the time. Some studies have shown that metal imagery activates the cortex through active mental simulation. Our previous study has shown that passive application of transcranial direct current stimulation causes subthreshold polarization and promotes the effective integration of residual brain high-level network. This study proposes a hypothesis: transcranial Direct Current Stimulation + Motor Imagery combines active and passive neuromodulation techniques to produce dual channel effect, which can synergistically excite motor cortex, remodel the motor network and optimize cerebral perfusion. The research contents include clarify the effect of transcranial Direct Current Stimulation + Motor Imagery neuromodulation therapy through comprehensive randomized controlled trial study; present the process of brain injury and secondary neural plasticity through the motor network construction, functional connectivity strength and cerebral perfusion with Blood Oxygen Level Dependent, Diffusion Tensor Imaging and Arterial Spin Labeling multimodal magnetic resonance technology; calculate the correlation between motor score and brain functional network, extract the key nodes that can promote the motor network remodeling. The research results are expected to provide preliminary theoretical foundations for further research on the injury and remodeling mechanism about upper extremity motor network after stroke.

ELIGIBILITY:
Inclusion Criteria:

* First stroke with upper limb motor dysfunction
* No rapid natural recovery in the last week
* Greater than 1 month since stroke onset
* Pass the motor imagery test

Exclusion Criteria:

* Severe cognitive disorder
* Severe spasm or joint contracture
* Mental implants in vivo
* Do not sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Behavioral assessment by Fugl-Meyer Assessment for Upper Limb | Baseline
  Complete the scale at baseline
Behavioral assessment by Fugl-Meyer Assessment for Upper Limb change | Immediately after intervention
  Change from baseline Action Research Arm Test immediately after intervention is obtained by subtracting the baseline from the later Fugl-Meyer Assessment score.
Behavioral assessment by Action Research Arm Test | Baseline
  Complete the above scale at baseline
Behavioral assessment by Action Research Arm Test change | Immediately after intervention
  Change from baseline Action Research Arm Test immediately after intervention is obtained by subtracting the baseline from the later Action Research Arm Test score.
Motor network construction | Baseline
  Construct the motor network with the bilateral primary motor cortices, supplementary motor cortices, premotor cortices, thalami and cerebellums et al. as the nodes of the network. Motor network analysis consists the network strength, global efficiency and local efficiency. The software used is PANDA and GRETNA.
Motor network change | Immediately after intervention
  Change from baseline motor network immediately after intervention is obtained by subtracting the baseline from the later network strength, global efficiency and local efficiency.
Cerebral perfusion calculation | Baseline
  The volume of interest covers the motor related territory including bilateral primary motor cortices, supplementary motor cortices, premotor cortices, thalami and cerebellums et al. The mean Cerebral Blood Flow value is calculated. The software used is Function Tool.
Cerebral perfusion change | Immediately after intervention
  Change from baseline cerebral perfusion immediately after intervention is obtained by subtracting the baseline from the later Cerebral Blood Flow value.

CONTACTS AND LOCATIONS:
Overall Officials: Lirong Huo, Doctor, Study Director — Office of academic research, Fu Xing Hospital, Capital Medical University
Locations (1):
- Fu Xing Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marquez JL, Conley AC, Karayanidis F, Miller J, Lagopoulos J, Parsons MW. Determining the benefits of transcranial direct current stimulation on functional upper limb movement in chronic stroke. Int J Rehabil Res. 2017 Jun;40(2):138-145. doi: 10.1097/MRR.0000000000000220. PMID 28196011
- [Background] Kaneko F, Shibata E, Hayami T, Nagahata K, Aoyama T. The association of motor imagery and kinesthetic illusion prolongs the effect of transcranial direct current stimulation on corticospinal tract excitability. J Neuroeng Rehabil. 2016 Apr 15;13:36. doi: 10.1186/s12984-016-0143-8. PMID 27079199
- [Background] Lioi G, Butet S, Fleury M, Bannier E, Lecuyer A, Bonan I, Barillot C. A Multi-Target Motor Imagery Training Using Bimodal EEG-fMRI Neurofeedback: A Pilot Study in Chronic Stroke Patients. Front Hum Neurosci. 2020 Feb 18;14:37. doi: 10.3389/fnhum.2020.00037. eCollection 2020. PMID 32132910
- [Background] Lee J, Lee A, Kim H, Shin M, Yun SM, Jung Y, Chang WH, Kim YH. Different Brain Connectivity between Responders and Nonresponders to Dual-Mode Noninvasive Brain Stimulation over Bilateral Primary Motor Cortices in Stroke Patients. Neural Plast. 2019 Apr 7;2019:3826495. doi: 10.1155/2019/3826495. eCollection 2019. PMID 31093270